CLINICAL TRIAL: NCT03480438
Title: Phase II Trial for the Treatment of Older Patients With Newly Diagnosed CD19 Positive, Ph/BCR-ABL Negative B-precursor Acute Lymphoblastic Leukemia With Sequential Dose Reduced Chemotherapy and Blinatumomab (EWALL-BOLD)
Brief Title: Treatment of Older Patients With B-precursor ALL With Sequential Dose Reduced Chemotherapy and Blinatumomab
Acronym: EWALL-BOLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, MD, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EWALL-BOLD
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: B-Precursor ALL
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Patients will receive blinatumomab at a dose of 28 μg/day as continuous intravenous infusion at constant flow rate for four weeks defined as one treatment cycle. Up to four cycles will be performed.
  In case of defined toxicities, the dose of blinatumomab may be reduced to 9 μg/day.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Patients will receive standard of care chemotherapy before blinatumomab, between blinatumomab cycles and after blinatumomab.
  Other Names: blincyto

SUMMARY:
The trial proposed here attempts to reduce induction chemotherapy to phase I of standard induction in patients with B-precursor ALL. Induction phase II will be replaced by blinatumomab.

The initial treatment phase is followed by sequential chemotherapy and further blinatumomab cycles.

DETAILED DESCRIPTION:
Blinatumomab is a bispecific single-chain antibody construct designed to link B cells and T cells resulting in T-cell activation and a cytotoxic T-cell response against CD19 expressing cells. In Phase II-III clinical trials 43-69 % of the patients treated with blinatumomab in relapsed/refractory ALL with poor prognostic features, achieved a complete hematologic remission and around 80 % of these obtained a molecular remission as well. Blinatumomab thus has demonstrated significant antileukemic activity in relapsed/refractory adult ALL. The ultimate goal for optimised management of adult ALL is to integrate targeted compounds with known single-drug activity into first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed CD19 positive B-precursor ALL
2. Greater than 25 % blasts in bone marrow
3. Eastern Cooperative Oncology Group (ECOG) performance status <= 2
4. Charlson comorbidity score <= 2
5. Age > 55 and < 75 years at the time of informed consent
6. Renal and hepatic function as defined below:

   * AST (SGOT), ALT(SGPT) and AP < 5x upper limit of normal (UNL) (unless related to leukemic liver infiltration by investigator assessment)
   * Total bilirubin < 1.5x ULN (unless related to Gilbert's Meulengracht disease)
   * Creatinine < 1.5x ULN
   * Creatinine clearance >= 50 mL/min (e.g. calculated according Cockroft & Gault)
7. Negative pregnancy test in women of childbearing potential
8. Ability to understand and willingness to sign a written informed consent
9. For Germany: Participation in the registry of the German Multicenter Study Group for Adult ALL (GMALL)

Exclusion Criteria:

1. Antileukemic pretreatment (GMALL prephase with dexamethasone and cyclophosphamide allowed)
2. History of malignancy other than ALL within 5 years prior to start of protocol-specified therapy with the exception of:

   * Malignancy treated with curative intent and with no known active disease present for 2 years before enrollment and felt to be at low risk for recurrence by the treating physician including
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated cervical carcinoma in situ without evidence of disease
   * Adequately treated breast ductal carcinoma in situ without evidence of disease
   * Prostatic intraepithelial neoplasia without evidence of prostate cancer
3. History or presence of clinically relevant (per investigator's assessment) CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or psychosis
4. Active ALL in the CNS confirmed by CSF analysis) or testes (clinical diagnosis) or other extramedullary involvement; non-bulky lymph node (< 7.5 cm diameter) involvement will be accepted
5. Current autoimmune disease or history of autoimmune disease with potential CNS involvement
6. Known exclusion criteria to recommended chemotherapy
7. Known positivity of HIV, hepatitis B (HbsAG) or hepatitis C virus (anti-HCV)
8. Subject received prior anti-CD19 therapy
9. Live vaccination within 2 weeks before the start of study treatment
10. Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation:

    Subject has known sensitivity to immunoglobulins or any of the products or components to be administered during dosing
11. Currently receiving treatment in another investigational device or drug study or less than 30 days since ending treatment on another investigational device or drug study(s). Thirty days is calculated from day 1 of protocol-specified therapy
12. Subject likely to not be available to complete all protocol-required study visits or procedures, including follow-up visits, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge
13. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety of interfere with the study evaluation, procedures or completion
14. Woman of childbearing potential and is not willing to use a highly effective method of contraception while receiving study treatment and for an additional 3 months after the last dose of study treatment
15. Male who has a female partner of childbearing potential, and is not willing to use 2 highly effective forms of contraception while receiving protocol-specified therapy and for at least an additional 3 months after the last dose of protocol-specified therapy.

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Hematologic and MRD response after induction therapy | after induction therapy (up to 8 weeks)
  Proportion of patients achieving a complete hematologic remission and a complete molecular remission (MRD response or complete MRD response) after induction therapy defined as one cycle of chemotherapy and one cycle of blinatumomab

SECONDARY OUTCOMES:
Overall Survival | 1 year after start of therapy
  Probability of overall survival at 1 year after start of therapy
Adverse Events | continuously until end-of-core-study (week 43)
  Rate and grade of adverse events (AE) according to CTC-AE in induction phase I, blinatumomab induction and during blinatumomab cycle I, II and III
MRD response after induction and consolidation | after induction and consolidation (up to 35 weeks)
  Proportion of patients who achieve a MRD response or a complete MRD response after induction consolidation
Time to MRD relapse | continuously until end of maintenance therapy (up to 27 months)
  Time to MRD relapse after prior achievement of MRD response or complete MRD response
Continuous complete remission | 1 year after start of therapy
  Probability of continuous complete remission at 1 year
Relapse free survival | 1 year after start of therapy
  Probability of relapse free survival at 1 year
Event-free survival | 1 year after start of therapy
  Probability of event-free survival at 1 year
Relapse localisation | In case of relapse, continuously until end of maintenance therapy (up to 27 months)
  Proportion of different relapse localisation in relation to total number of relapses
Quality of life | until end of maintenance therapy (up to 27 months)
  Quality of life measures (EORTC=European Organisation for Research and Treatment of Cancer standard scales) at different time-points during induction and consolidation; this is a multidimensional questionnaire with different scales per item such als functional scale, global health status and symptoms. Details are outlined in respective manuals (https://qol.eortc.org/manuals/)
Treatment deviation 1 | until end of treatment (up to 39 weeks)
  Rate of treatment interruptions
Treatment deviation 2 | until end of treatment (up to 39 weeks)
  Duration of treatment interruptions
Treatment deviation 3 | until end of treatment (up to 39 weeks)
  Dose reductions
Treatment deviation 4 | until end of treatment (up to 39 weeks)
  Mitigation strategies
Treatment deviation 5 | until end of treatment (up to 39 weeks)
  Rate of withdrawals

OTHER OUTCOMES:
Hospitalisation time | until end of treatment (up to 39 weeks)
  Number of hospitalisation days
Infusion pump systems | until end of treatment (up to 39 weeks)
  Use of infusion pump systems
Ambulatory care services | until end of treatment (up to 39 weeks)
  Use of ambulatory care services
Biologic markers | continuously until end of consolidation therapy (up to 35 weeks)
  Measurement of biologic markers in bone marrow and peripheral blood throughout induction and consolidation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, MD, Study Director — Johann Wolfgang Goethe University Hospital
Locations (21):
- Germany (21):
  - University Hospital of Frankfurt (Main), Frankfurt am Main, Hesse
  - Uniklinik RWTH Aachen, Aachen
  - Charité - Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen Mitte, Bremen
  - Evangelisches Krankenhaus Essen-Werden, Essen
  - Universitätsklinikum Halle, Halle
  - Uniklinik Hamburg Eppendorf, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Gemeinschaftsklinikum Mittelrhein, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Großhadern, München
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Helios Klinikum Wuppertal, Wuppertal
  - Uniklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial register of the Kompetenznetz Leukaemie — https://www.kompetenznetz-leukaemie.de
- See also: Clinical Trials Register Results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-002853-13/results